CLINICAL TRIAL: NCT00394485
Title: A Randomized Crossover Trial Comparing the Efficacy and Safety of Tiotropium + Procaterol vs. Tiotropium + Placebo in Moderate COPD Patients
Brief Title: Tiotropium + Procaterol vs Tiotropium + Placebo in COPD Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficulty in recruting patients
Sponsor: Otsuka Pharmaceutical, Inc., Philippines (Industry)
Collaborators: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Co, Benjamin, Medical Director, Otsuka Pharmaceutical, Inc., Philippines
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: OPPI-MPTA-COPD-1
Record Dates: First submitted 2006-10-31; First posted 2006-11-01 (Estimated); Last update posted 2009-12-17 (Estimated); Status verified 2009-12

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Chronic Obstructive Pulmonary Disease; Procaterol; Tiotropium
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Procaterol; Tiotropium Bromide

INTERVENTIONS:
Drug: Procaterol
Drug: Tiotropium

SUMMARY:
Study compares the efficacy and safety of tiotropium + a beta agonist (procaterol) vs. tiotropium alone among patients with moderate chronic obstructive pulmonary disease

DETAILED DESCRIPTION:
This study aims to determine the efficacy and safety of tiotropium plus procaterol in comparison to tiotropium plus placebo in Filipino patients seen in Manila, with moderate COPD.

After a 1-week wash-out period, 6-minute walk test, and St. George's Respiratory Questionnaire (SGRQ) will then be administered prior to a run-in period of 1 week wherein all patients will be started on tiotropium alone. The patients will then be randomly allocated to either of the two arms for a two-week treatment, followed by one week washout, and crossed-over to the other treatment for another two weeks. The procaterol or placebo dose is given 2 hrs after the tiotropium dose.

ELIGIBILITY:
Inclusion Criteria:

1. GOLD criteria for moderate COPD (post-bronchodilator)

   * FEV1/FVC < 70%
   * 50% ≤ FEV1 < 80% predicted
   * With or without symptoms
2. Willing to undergo the treatment protocol with signed informed consent

Exclusion Criteria:

1. Exacerbation within 1 month prior to run-in period
2. Significant hypoxemia and/or desaturation at rest and during exercise.
3. Significant cardiac, renal, or other systemic disease
4. History of adverse reaction to any of the two test drugs (tiotropium and procaterol)

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2006-05; Study Completion 2008-04

PRIMARY OUTCOMES:
[Efficacy] Improvement spirometry (FEV1, FVC, FEV1/FVC, 6 MWD, TDI) and SGRQ at 2 weeks

SECONDARY OUTCOMES:
[Safety] HR (Heart Rate) and BP (Blood Pressure)
Incidence of adverse reactions and changes

CONTACTS AND LOCATIONS:
Overall Officials: Abundio A Balgos, MD, Principal Investigator — University of the Philippines College of Medicine
Locations (1):
- Philippine General Hospital, Manila, National Capital Region, Philippines